CLINICAL TRIAL: NCT04169230
Title: The Effect of Acute Citalopram on Self-referential Emotional Processing and Social Cognition in Healthy Volunteers
Brief Title: Citalopram and Self Emotional Processing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: University of Bath (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Acute_Citalopram
Record Dates: First submitted 2019-11-12; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Molecular Mechanisms of Pharmacological Action; Depression; Depressive Disorder; Mental Disorder; Antidepressive Agents; Cognition
Keywords: Citalopram; Emotional Processing; Antidepressants; Self Processing; Healthy Volunteers
MeSH Terms: conditions — Depression; Depressive Disorder; Mental Disorders | interventions — Citalopram

STUDY DESIGN:
Intervention Model Description: Following the screening, eligible participants will be randomised to receive either a single 20mg oral dose of citalopram or a matched lactose placebo tablet using an online randomisation tool. Note that the study is not assessing the safety or efficacy of citalopram, but rather using it as a probe to understand the role of serotonin in self-referential emotional processing biases.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citalopram (Experimental): Single acute oral dose 20 mg Citalopram (tablet encapsulated in opaque capsule)
  Interventions: Drug: Citalopram
- Placebo (Placebo Comparator): Single acute oral dose Lactose Placebo (tablet encapsulated in opaque capsule)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Citalopram — Single dose administration of citalopram (20mg)
  Arms: Citalopram
Drug: Placebo oral tablet — Single dose administration lactose placebo tablet
  Arms: Placebo

SUMMARY:
This study is investigating the effect of an acute dose of citalopram on emotional processing about the self. Using a parallel-group double-blind design, participants will be randomised to receive either an acute dose of citalopram or placebo. Participants will then complete a number of widely used computer-based cognitive tasks measuring emotional processing biases towards the self.

This study has also been registered on OSF: https://osf.io/nhjvs/?view_only=b39c49bddfd543b99b627dc992e49b45

DETAILED DESCRIPTION:
Antidepressants are thought to operate by changing the way patients process emotional information. After a single dose of citalopram or fluoxetine healthy volunteers have been found to display an increased recognition of happy facial expressions and a reduced recognition of sad faces, in the absence of changes in mood. Studies using depressed participants have produced similar results. However, there has been comparatively little research on changes in emotional processing biases about the self following antidepressant administration. Sense of self has been proposed as fundamental for mental health, with self-schemas acting as a focus through which valence and reward influenced perception, memory and decision-making. Antidepressants may increase learning of positive information about the self, potentially remediating negative self-schema and subsequently reducing depression symptoms.

In this study, the investigators aim to examine whether acute administration of citalopram is associated with an increase in positive emotional learning biases about the self. Using a parallel-group double-blind design, participants will be randomised to receive either an acute dose of citalopram or placebo. Participants will then complete a number of widely used computer-based cognitive tasks measuring emotional processing biases. Identifying early changes in cognition and behaviour following antidepressant treatment will increase our knowledge of how antidepressants operate, and provide putative targets to identify early response to antidepressants.

This study has also been registered on OSF: https://osf.io/nhjvs/?view_only=b39c49bddfd543b99b627dc992e49b45

Starting from the 8th November 2019 an additional task (the Oxford Cognition Stress Task (OCST)) was included in the test battery. This task has been developed by the Psychopharmacology and Emotion Research Laboratory (PERL), Department of Psychiatry, University of Oxford. This is an acute psychosocial stress induction paradigm, comprised of computerised cognitive tasks with an induced failure component. An algorithm varies task timing/difficulty to be just beyond participants' ability, accompanied by aversive feedback. The OCST induces mild, transient increases in stress and arousal, as indexed by heart rate, skin conductance, salivary cortisol and self-reported subjective state measures. Data for this task will be collected, analysed and published by PERL and will not be included in any publications relating to the previous registration for this study. The OCST task has been included at the end of the test battery and is therefore not expected to influence data relating to any self-report measures or tasks outlined in the previous registration

This section of the study has been registered separately on ClinicalTrials.gov (titled 'Citalopram and Stress Reactivity') to reflect the separate research questions and study team involvement.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Aged 18 -45 years
* Fluent in written and spoken English at a sufficient level to understand and complete the tasks
* Body Mass Index (BMI) 18-30
* Participant is willing and able to give informed consent for participation in the study
* Not currently taking any regular medications (expect the contraceptive pill)

Exclusion Criteria:

* Any past or current Axis 1 DSM-V psychiatric disorder
* Current use of psychoactive medication (except the contraceptive pill, the Depo-Provera injection or the progesterone implant)
* Current or past history of drug or alcohol dependency
* History of current significant neurological condition (e.g. epilepsy)
* Known hypersensitivity to the study drug
* Currently pregnant or breast feeding
* Previous participation in a study that uses the same or similar computer tasks as those used in the present study
* Previous participation in a study that involves the use of a medication within the last three months
* Significant medical condition
* Smokers consuming > 5 cigarettes per day
* Individuals consuming > 6 caffeinated drinks per day
* Lactose Intolerance (due to the study involving administration of a lactose placebo tablet)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Social Evaluation Learning Task: Bias Scores | Day 1: 3-5.5 hours post drug administration
  An overall index of positive or negative bias will be calculated for each referential condition (self, friend, stranger) using errors to criterion (the number of errors made before 8 rule-congruent responses). Bias is calculated by subtracting errors to criterion made when learning the dislike rule from errors to criterion made when learning the like rule. A positive value indicates a negative bias, as fewer errors are made learning the dislike rule compared to the like rule. Conversely, a negative value indicates a positive bias, as fewer errors are made learning the like rule compared to the dislike rule. The minimum possible value is - 24 (complete bias towards being liked), and the maximum value is + 24 (complete bias towards being disliked).
Associative Learning Task: Reaction Times (ms) | Day 1: 3-5.5 hours post drug administration
  Mean reaction times will be calculated for each referential condition (self, friend, stranger), reward condition (high, medium, low) and valence condition (positive, neutral, negative) for each respective task.
Associative Learning Task: Accuracy (% correct) | Day 1: 3-5.5 hours post drug administration
  Mean accuracy will be calculated for each referential condition (self, friend, stranger), reward condition (high, medium, low) and valence condition (positive, neutral, negative) for each respective task.
Self-Esteem Go/No-Go Association Task: d' | Day 1: 3-5.5 hours post drug administration
  Discriminative accuracy (d') will be calculated through applying Z-score transformations, and subtracting hit z-scores from false alarm z-scores. Z-scores are adjusted by adding or subtracting .005 if hit or false-alarm rates are 0 or 1. d' -values can then be compared for each possible categorical combination to examine implicit self-biases.

SECONDARY OUTCOMES:
Prisoner's Dilemma: Cooperative Behaviours (%) | Day 1: 3-5.5 hours post drug administration
  The main outcome for this task is the proportion of rounds on which participants choose to cooperate. The conditional probability of cooperating will be calculated according to the proportion of rounds on which participants cooperated following each of the four possible outcomes.
Prisoner's Dilemma: Reaction Times (ms) | Day 1: 3-5.5 hours post drug administration
  Reaction times for cooperation versus non-cooperation choices will be calculated.
Emotional Categorisation and Recall: Number of words categorised | Day 1: 3-5.5 hours post drug administration
  The mean number of positive and negative words categorised as describing or not describing the participant/the other will be recorded.
Emotional Categorisation and Recall: Hits | Day 1: 3-5.5 hours post drug administration
  Mean hits will be collected for each referential condition and valence.
Emotional Categorisation and Recall: False Alarms | Day 1: 3-5.5 hours post drug administration
  Mean alse intrusions will be collected for each referential condition and valence.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Harmer, DPhil, Principal Investigator — University of Oxford; Katherine S Button, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised dataset will be published as open access data on a secure online repository, such as Open Science Framework (https://osf.io/). Participant IDs will be randomly reassigned in this dataset to ensure complete removal of any linkage between anonymised and personal data. Self-report questionnaire data and task outcomes will be included.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: An anonymised dataset will be shared after full anonymisation of study data and publication of findings. Data will be available indefinitely.

REFERENCES:
- See also: PERL Oxford — https://www.psych.ox.ac.uk/research/psychopharmacology-and-emotion-research-laboratory

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT04169230/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT04169230/ICF_001.pdf